CLINICAL TRIAL: NCT07304310
Title: Clinical Evaluation of Two Minimally Invasive Protocols for Orthodontic Clean-Up: A Case-Control Study
Brief Title: Comparison of Two Orthodontic Clean-Up Protocols
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Simona Tecco, Associate Professor, IRCCS San Raffaele
Other Study IDs: OCUs
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Orthodontic Appliance; Debonding; Case-control Study
Keywords: orthodontic clean-up; orthodontic debonding; enamel preservation; minimally invasive dentistry; case-control study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients underwent orthodontic clean-up with a two-step ultrasonic system (Combi Touch, Mectron) equipped with 30-µm diamond-coated and PEEK-coated inserts
  Interventions: Device: Two-step ultrasonic protocol
- Control group: Patients underwent orthodontic clean-up with a one-step tungsten carbide/abrasive polisher (One Gloss®, Shofu)
  Interventions: Device: One-step clean-up protocol

INTERVENTIONS:
Device: Two-step ultrasonic protocol — Diamond- and PEEK-coated inserts
  Groups: Case group
Device: One-step clean-up protocol — One-step tungsten carbide/abrasive polisher
  Groups: Control group

SUMMARY:
Orthodontic clean-up following debonding remains a technically demanding procedure, with documented risks of enamel roughening, microdefects, discoloration, and increased plaque retention. Minimally invasive technologies have recently been introduced to improve adhesive removal while limiting damage to the outer enamel layer, but comparative clinical evidence remains limited. This aim of this case-control study was to compare the effectiveness and the safety of two different minimally invasive clean-up systems: two-step ultrasonic inserts (Combi Touch, Mectron) and a one-step polishing bur (One Gloss®, Shofu).

A total of 142 patients presenting residual orthodontic adhesive after debonding were included. They were randomly allocated to: (1) Case group (n = 71): two-step ultrasonic system (Combi Touch, Mectron) equipped with 30-µm diamond-coated and PEEK-coated inserts; (2) Control group (n= 71): one-step tungsten carbide/abrasive polisher (One Gloss®, Shofu). For each patient the following clinical indices were recorded at baseline (T0) and 30-day follow-up (T1): Plaque Control Record (PCR), Bleeding on Probing (BoP), Adhesive Remnant Index (ARI), International Caries Detection and Assessment System (ICDAS-II), and dentinal sensitivity (Schiff Air Index). Orthodontic treatment modality (clear aligners vs fixed appliances) was documented as a covariate and tested for potential interactions with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone either fixed vestibular orthodontic treatment or clear aligner therapy
* Debonding procedure must not have occurred more than 24 months prior to evaluation
* ICDAS-II index ≤ 2

Exclusion Criteria:

* Patients treated with removable orthodontic appliances
* Patients whose debonding exceeded 24 months
* ICDAS-II score > 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of 142 consecutive patients requiring adhesive removal following orthodontic debonding. Participants were recruited at the Oral Hygiene and Prevention Center of the Department of Dentistry, San Raffaele Hospital, and at the Smart Dental Clinics (San Donato Group), Milan, Italy, between April 2025 and September 2025.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Plaque Control Record (PCR) | Baseline, after 30 days
  The PCR is scored as the percentage of tooth surfaces with visible plaque (0-100%). Higher scores indicate worse oral hygiene.
Bleeding on Probing (BoP) | Baseline, after 30 days
  BoP is expressed as the percentage of bleeding sites (0-100%). Higher scores indicate worse gingival health.
Adhesive Remnant Index (ARI) | Baseline, after 30 days
  The ARI is scored 0-3, where 0 = no adhesive left on tooth surface and 3 = all adhesive remaining. Higher scores indicate more adhesive remaining on the enamel.
International Caries Detection and Assessment System (ICDAS-II) | Baseline, after 30 days
  The ICDAS-II is scored from 0 to 6, where 0 = sound tooth surface and 6 = extensive cavitated lesion. Higher scores indicate worse caries status.
Schiff Air Index | Baseline, after 30 days
  The Schiff Air Index scored from 0 to 3, where 0 = no response to air stimulus and 3 = strong painful response. Higher scores indicate greater dentinal hypersensitivity.

SECONDARY OUTCOMES:
Orthodontic treatment modality | Baseline
  Orthodontic treatment modality was recorded as a categorical variable at baseline (T0), distinguishing between the use of clear aligners and fixed appliances. This variable does not follow a numerical scale; instead, it consists of two categories. No minimum or maximum values apply, and higher values do not correspond to better or worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic, IRCCS San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pont HB, Ozcan M, Bagis B, Ren Y. Loss of surface enamel after bracket debonding: an in-vivo and ex-vivo evaluation. Am J Orthod Dentofacial Orthop. 2010 Oct;138(4):387.e1-387.e9. doi: 10.1016/j.ajodo.2010.01.028. PMID 20889035
- [Background] D'Amario M, Bernardi S, Di Lauro D, Marzo G, Macchiarelli G, Capogreco M. Debonding and Clean-Up in Orthodontics: Evaluation of Different Techniques and Micro-Morphological Aspects of the Enamel Surface. Dent J (Basel). 2020 Jun 17;8(2):58. doi: 10.3390/dj8020058. PMID 32560482
- [Background] Thawaba AA, Albelasy NF, Elsherbini AM, Hafez AM. Evaluation of enamel roughness after orthodontic debonding and clean-up procedures using zirconia, tungsten carbide, and white stone burs: an in vitro study. BMC Oral Health. 2023 Jul 13;23(1):478. doi: 10.1186/s12903-023-03194-6. PMID 37443027
- [Background] Campbell PM. Enamel surfaces after orthodontic bracket debonding. Angle Orthod. 1995;65(2):103-10. doi: 10.1043/0003-3219(1995)0652.0.CO;2. PMID 7785800